CLINICAL TRIAL: NCT05436873
Title: Evaluation of Sonalleve MR-HIFU for Non-invasive Thermal Therapy of Facet-Joint Syndrome: Feasibility and Safety Clinical Study
Brief Title: MR-HIFU for Non-invasive Thermal Therapy of Facet-Joint Syndrome:
Acronym: HIFU-FACET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Uni-Koeln-4473
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Facet Joint Syndrome

STUDY DESIGN:
Intervention Model Description: There is only 1 treatment arm, as this is a feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): This is a single arm study
  Interventions: Device: MR-HIFU

INTERVENTIONS:
Device: MR-HIFU — MRI guided High Intensity Focused Ultrasound sonication.

SUMMARY:
Patients suffering from facet-joint-syndrome associated with lower-back pain will be treated with MRI-guided High Intensity Focused Ultrasound thermal therapy for pain relief.

DETAILED DESCRIPTION:
Patients with diagnosed facet-joint-syndrome are suffering from severe pain in the respective regions, mainly lower-back pain. Eligible patients will be treated with High Intensity Focused Ultrasound (HIFU) under MRI control. The control by MRI assures on the one hand the correct selection of area to be sonicated and monitors in parallel the temperature, reached in the target area. The aim is to thermally ablate facet joint and/or medial branch nerves at lumbar spine. Ablation is deemed to be feasible and successful if temperatures of at least 57°C are reached at the target. The entire procedure will be done under anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain
* clinical diagnosis of Lumbar Facet Joint Syndrome
* eligible for MRI and MR-HIFU session
* eligible for general anaesthesia
* intact skin and soft tissue over treatment zone
* facet joint anatomy clearly identifiable
* patients must be able to discontinue all pain relief medication for a minimum of 48 hours prior to baseline assessment
* patients able to provide consent for the study

Exclusion Criteria:

* spinal implants
* treatment target zone < 10 mm from the skin
* pregnant female patients
* breastfeeding female patients
* body weight > 140 kg
* systemic and/or local infections
* moderate to high grade of spinal instability
* MRI contrast agent contraindication
* any MRI-unsafe implant or pacemaker
* facet joint anatomy which is not targetable or reachable due to scars, surgical clips, implants, or prosthesis in the planned beam path of the ultrasound beam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility: planned temperature (57°C) achieved at target area of sonication | treatment day (4 hours)
  Temperatures achieved at the intended treatment location during MR-HIFU treatments

SECONDARY OUTCOMES:
safety of entire procedure | 180 days
  Frequency and severity of adverse events associated with use of the Sonalleve MR-HIFU system
Pain reduction after study treatment | 180 days
  pain reduction as shown in VAS and change in frequency/type/dosing of pain relief medication
change in Quality of Life (QoL) assessed via Quality of Life Questionnaire | 180 days
  The change in QoL scores throughout study participation [as higher values, as better quality of Life]
comparison of contrast in MRI before and after treatment | 180 days
  Qualitative analysis of the change in image tissue contrast in MRI images taken prior, during and after the treatment. This is a visual evaluation only.

CONTACTS AND LOCATIONS:
Overall Officials: Kourosh Zarghooni, PD, Principal Investigator — Department of Orthopaedics and Trauma Surgery; Cologne University Hospital; Kerpener Strasse 62; D 50937 Cologne
Locations (1):
- Holger Gruell, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided